CLINICAL TRIAL: NCT00491374
Title: A Double-Blind Placebo-Controlled, Randomized, Parallel-Group, Single-Site Study Of Mometasone Furoate Nasal Spray (MFNS) In Subjects With Mild-Moderate Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) Associated With Perennial Allergic Rhinitis (PAR) Using Polysomnographic Recordings of Sleep Parameters
Brief Title: Study of Nasonex® in Improving Sleep Disturbances Related to Perennial Allergic Rhinitis (Study P04909)(TERMINATED)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Very poor enrollment
Sponsor: Schering-Plough (Industry)
Responsible Party: Head, Clinical Trials Registry & Results Disclosure Group, Schering-Plough
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04909
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Results first posted 2009-01-06 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MFNS (Experimental)
  Interventions: Drug: Mometasone Furoate Nasal Spray
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray — Nasonex Nasal Spray 50 mcg/spray, 200 mcg (4 sprays) once daily every morning for 28 days.
  Other Names: SCH 32088
  Arms: MFNS
Drug: Placebo — Placebo Nasal Spray 4 sprays once daily every morning for 28 days.
  Arms: Placebo

SUMMARY:
This study will hope to show that the treatment of the patient's perennial allergic rhinitis (PAR) using Nasonex® (mometasone furoate nasal spray) will result in improvement of the nasal symptoms of PAR and of nighttime sleep-disordered breathing, thereby resulting in improved sleep quality, less daytime sleepiness, improved daytime functioning, and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 to 45 years of age, of either sex, and any race.
2. Must have at least a 2-year history of PAR.
3. Must be skin test positive for the usual allergens associated with PAR within the previous 12 months with regular exposure to at least one of the allergens to which the subject is allergic.
4. Must be sufficiently symptomatic at the Screening Visit (Visit 1), Qualification Visit (Visit 2), and Baseline Visit (Visit 4) with a minimal level of PRIOR (reflective) total symptom score, total nasal symptoms score, and total non-nasal symptoms score in order to qualify.
5. At the Qualification Visit 2, subjects must have a score of at least 2 with the Interference with Sleep severity rating score for at least 3 of the 7 nights prior to the Qualification visit.
6. At the Baseline Visit 4 subjects must have a score of at least 2 with the Interference with Sleep severity rating score for at least 1 of the 3 nights prior to the Baseline Visit.
7. Must have an apnea-hypopnea index (AHI) of >=5, but not more than 30, during the first screening polysomnographic evaluation and to proceed to the second polysomnographic evaluation.
8. At the Baseline Visit (Visit 4), the subjects must complete the NRQLQ, PQSI, ESS, WPAI-AS.
9. Must complete the PVT within 1 hour of bedtime and 1 hour of arising on the nights when the PSGs are done.
10. Female subjects of childbearing potential (including women who are less than 1 year postmenopausal and women who will be sexually active during the study) must agree to use a medically accepted method of contraception or be surgically sterilized prior to screening, while receiving protocol-specified medication, and for 30 days after stopping the medication. Women who are postmenopausal for >1 year (ie, women who have experienced 12 consecutive months of amenorrhea) will be exempted from the use of contraception during the study.
11. Female subjects of childbearing potential must have a negative urine pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Visit 4 confirmed prior to dosing with the study drug and at final Visit 7.

Exclusion Criteria:

1. Subject has symptomatic seasonal allergic rhinitis (SAR) or a history of SAR during the same calendar period as this study.
2. Subject is a female who is pregnant, or intends to become pregnant during the study.
3. Subject is nursing, or intends to be nursing during the study.
4. Subject has used any investigational product within 30 days prior to enrollment or any antibodies for asthma or allergic rhinitis in the past 90 days).
5. Subject has any of the following clinical conditions:

   * known severe sleep apnea
   * asthma
   * chronic obstructive pulmonary disease (COPD)
   * alcohol abuse
   * rhinitis medicamentosa
6. Subject is currently on or has been on an antihistamine, decongestant (topical or systemic) or a nasal inhaled corticosteroid during the 14 days prior to the Screening Visit.
7. Subject with current or history of frequent episodes (2 or more episodes per year for the past 2 years) of clinically significant sinusitis or chronic purulent postnasal drip.
8. Subject has had recent nasal septum ulcers, nasal surgery, or nasal trauma.
9. Subject has had an upper or lower respiratory tract or sinus infection that required antibiotic therapy with the last dose 14 days prior to screening, or who has had a viral upper or lower respiratory infection within 14 days prior to screening.
10. Subject has nasal structural abnormalities, including large nasal polyps, and marked septum deviation that significantly interfere with nasal airflow.
11. Subject is unable to refrain from regular use of nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids.
12. Subject on immunotherapy (desensitization therapy) should not receive an increase in dose during the study. Subjects may not receive desensitization treatment within 24 hours prior to a study visit.
13. Subject has active or quiescent tuberculosis infection of the respiratory tract, untreated fungal, bacterial, or systemic viral infections, or ocular herpes simplex.
14. Subject is morbidly obese (BMI >=35).
15. Subject is a night-shift worker and does not have a standard asleep at night / awake during the day cycle, or has an irregular sleep/wake schedule.
16. Subject reports routinely spending less than 6 1/2 hours of time in bed per night.
17. Subject reports drinking 3 or more cups of regular coffee or 4 or more 8 ounce cans/bottles of caffeine-containing carbonated beverages per 24 hour period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Study Completion 2007-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No subject fulfilled the requirements for randomized assignment of treatment; thus, no subject was assigned an intervention, and no subject was treated. The trial was terminated.
Period: Overall Study
Arm/Group | Placebo | Mometasone Furoate Nasal Spray
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mometasone Furoate Nasal Spray | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Customized [Number; unit: participants]
  Any Age | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Either Sex | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in the Number of Apnea-hypopnea Episodes Per Hour (Apnea-hypopnea Index (AHI)
Population: The primary outcome measure could not be assessed because no subject received randomized treatment assignment, or any treatment. The study was terminated.
Measure: Number
Arm/Group | Placebo | Mometasone Furoate Nasal Spray
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Mometasone Furoate Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0 | 0
Other Adverse Events (participants affected / at risk) | 0 | 0

LIMITATIONS AND CAVEATS:
This study was difficult to enroll subjects, and after 5 months of screening, the screen failure rate was 100%. At that time the decision was made to terminate the study. No subject was treated and no data were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other